CLINICAL TRIAL: NCT03802136
Title: Prognostic Value of Early Oxidative Stress Biomarkers in Patients With Sepsis
Brief Title: Multiple Biomarkers in ICU Sepsis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, ZhiYong Peng, professor, Zhongnan Hospital
Other Study IDs: 2018062
Record Dates: First submitted 2019-01-02; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Sepsis, Severe; Sepsis; Septic Shock; AKI
Keywords: AKI; Sepsis; Biomarker; renal function; oxidative stress
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and centrifuged urine will be retained in a -80℃ fridge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high concentration of biomarkers: the patients with biomarkers level over the normal max value
- low concentration of biomarkers: the patients with biomarkers level below the normal max value

SUMMARY:
Acute kidney injury (AKI) is a common condition among sepsis patients in the intensive care unit (ICU) and is associated with high morbidity and mortality. Oxidative stress biomarkers were investigated in panels and were reported to predict renal failure in sepsis patients. Some biomarkers would be able to identify who will recover and not recover better than serum creatinine. Thus, a combining oxidative stress biomarkers are needed to predict the occurrence or progression of AKI in critically ill patients.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common condition among sepsis patients in the intensive care unit (ICU) and is associated with high morbidity and mortality. Oxidative stress biomarkers were investigated in panels and were reported to predict renal failure in sepsis patients. Research on AKI has focused on new damage biomarkers for early detection of AKI and worsening of renal function. Some biomarkers would be able to identify who will recover and not recover better than serum creatinine. Thus, a combining functional and damage markers as well as oxidative stress biomarkers are needed to predict the occurrence or progression of AKI in critically ill patients. Therefore, this prospective, observational study will be conducted in Mainland China

ELIGIBILITY:
Inclusion Criteria:

* sepsis patients in appropriate age

Exclusion Criteria:

* ever blood transfusion ever CPR（cardiopulmonary resuscitation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to ICU of Zhongnan Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-30 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
presence of AKI | a week after admission to ICU
  Use serum creatinine or urine output（The KDIGO Guidelines 2012) to asess whether AKI happens to the studied subjects within a week after admission to ICU
Death of the patients | 2 weeks after admission to ICU
  Mortality of the studied patients

SECONDARY OUTCOMES:
Use serum creatinine to assess renal function of the patients | the 1 day when the patients admitted to ICU
  Concetration of serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: zhiyong peng, professor, Study Director — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China